CLINICAL TRIAL: NCT01832077
Title: The Impact of Telemedicine System to the Diagnosis and Treatment of Diabetes Retinopathy in Rural Canton
Brief Title: Uptake of Telemedicine System Trial in Rual Canton
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Collaborators: Orbis (Other); The World Diabetes Foundation (Other)
Responsible Party: Principal Investigator, Congdon Nathan, vice director,Blindness Prevention and Treatment Department, Sun Yat-sen University
Other Study IDs: ZOC-WDF-Telemedicine
Record Dates: First submitted 2013-04-11; First posted 2013-04-15 (Estimated); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Diabetes Retinopathy; Diabetes Macular Edema
Keywords: sensibility; specificity; positive predictive value; negative predictive value; Cost-effectiveness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- rural doctor: examine patient's fundus by 90D fundus pre-set lens
  Interventions: Device: 90 D
- grader: grade fundus pictures in ZOC
  Interventions: Device: fundus camera and grader

INTERVENTIONS:
Device: 90 D — rural doctors exam eye fundus by 90 D
  Groups: rural doctor
Device: fundus camera and grader — taking fundus pictures and graded by graders in ZOC
  Groups: grader

SUMMARY:
To evaluate the impact of telemedicine system in rural hospitals for diagnosis and treatment of Diabetes retinopathy and Diabetes macular edema.

DETAILED DESCRIPTION:
Telemedicine system mainly contains a comprehensive eye examination electric-records (E-record), which can transfer the fundus pictures from rural hospitals to professional Graders (golden standard for a diagnose of Diabetes Retinopathy (DR) and Diabetes Macular Edema(DME)). In Zhongshan Ophthalmic Center (ZOC). By this system, the investigators can evaluate the capacity of rural eye doctors about the diagnosis of DR/DME, and give proper suggestions for the treatment and revisit plan.

ELIGIBILITY:
Inclusion Criteria:

* age > 40y, diagnosed (Diabetes Retinopathy) DR,10% normal patients

Exclusion Criteria:

* unconsciousness, history of diabetic ketoacidosis, cardiac insufficiency, Severe atrioventricular block, hepatic insufficiency , allergic to mydriatic

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: age > 40y, diagnosed (Diabetes Retinapathy)DR, 10% normal patients
Sampling Method: Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Accuracy of trained doctors in diagnosing DR/DME versus photo grading and automated grading | 2 years after the telemedicine begin to use
  To compare the sensitivity, specificity and positive and negative predictive value for a diagnosis of DR/DME , a diagnosis of DR/DME requiring treatment, of trained rural doctors and an automated grading system, as compared to trained graders using photographs (the gold standard)
cost-effectiveness | 2 years
  Cost-effectiveness of three methods of DR screening (trained rural doctors versus telemedicine versus automated grading)

SECONDARY OUTCOMES:
Frequency of comprehensive eye examination taken by rural doctors | 2 years
  Frequency with which trained rural doctors continue to implement suggested examinations (IOP, gonioscopy, pupil exam, dilated examination)
comprehensive eye examination rate among patients in rural hospitals | 2 years
  Frequency with which patients get comprehensive eye examinations in rural hospitals, and its influencing factors.
the usage rate of Electric-Record | 2 years
  to evaluate the usage rate of E-record by rural doctors when they see patients in the eye clinic, and its influencing factors.
Cost-effectiveness of van | 2 years
  compare the cost-effectiveness of van for laser treatment to DR/DME patients with the transfer treatment in ZOC

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Congdong, MD,MPH, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, No.54, Xianlienan Road, Guangzhou, Guangdong, China